CLINICAL TRIAL: NCT00585871
Title: Clonidine to Prevent Implantable Cardiovertor Defibrillator Firing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: could not recruit
Sponsor: James Martins (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, James Martins, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200602703; study is over no ID is needed
Record Dates: First submitted 2007-12-29; First posted 2008-01-03 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Ventricular Tachycardia
Keywords: ICD patients with 5 VTs per 3 month period
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Clonidine; Metoprolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clonidine therapy group (Experimental): clonidine 0.1 TID
  Interventions: Drug: clonidine
- Metoprolol control group (Active Comparator): metoprolol 25 TID
  Interventions: Drug: metoprolol

INTERVENTIONS:
Drug: clonidine — 0.1 mg tid
  Arms: Clonidine therapy group
Drug: metoprolol — 25 mg tid
  Arms: Metoprolol control group

SUMMARY:
Cardiac arrest or sustained VT (ventricular tachycardia) in patients with heart disease is best treated with an ICD (implantable cardioverter defibrillator). However, the ICD alone is not appropriate therapy for patients with frequent VT episodes. In fact frequent shocks for VT may predict a poorer prognosis. Anti-arrhythmic drugs are co-administered with ICDs in up to 50% of patients to prevent VT episodes, but antiarrhythmic drugs may have harmful effects. Thus improved drugs to prevent VT without interfering with ICD function are needed. Recent data including our own suggest that clonidine may be a new therapy to prevent ICD shocks. It may act centrally on sympathetic outflow and peripherally and selectively on cardiac Purkinje, to suppress and control VT occurring in patients. Our purpose is to test the hypothesis that clonidine reduces frequent VT better than beta blocker in patients with ICDs. After informed consent patients will be randomized in a single blind fashion to either clonidine or metoprolol given three times per day. Other prescribed drugs may be adjusted to promote toleration of the study drug. ICD interrogations of episodes of VT will be the primary endpoint. Device based NIPS (non-invasive programmed stimulation) testing in a subset of these patients will allow mechanistic understanding of the clonidine effect. All of the procedural techniques are in place as performed clinically; preliminary data are given showing feasibility of the project.

DETAILED DESCRIPTION:
we had wanted very commonly occurring VT episodes on ICD interrogation: 5 episodes/ 3 months. We could not enroll more than 2 patients most of which have interventions to prevent episodes. Thus we could not enroll patients and discontinued the study in the first year.

ELIGIBILITY:
Inclusion Criteria:

* Implantable defibrillator treated patients with 5 episodes of ventricular tachycardia per 3 month period

Exclusion Criteria:

* No more than one shock/3 months
* No contraindication to clonidine
* Non-compliance
* Asthma

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
episodes of non-sustained ventricular tachycardia | one year

SECONDARY OUTCOMES:
defibrillator shocks | one year

CONTACTS AND LOCATIONS:
Overall Officials: james b martins, md, Principal Investigator — University of Iowa
Locations (1):
- UIHC, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No